CLINICAL TRIAL: NCT03729544
Title: Randomized Controlled Trial of Electronic Alert-Based Computerized Decision Support to Increase Detection of Chronic Thromboembolic Pulmonary Hypertension in Patients With Prior Pulmonary Embolism (CTEPH-DETECT)
Brief Title: Computerized Decision Support to Increase Detection of Chronic Thromboembolic Pulmonary Hypertension in Patients With Prior Pulmonary Embolism
Acronym: CTEPH-DETECT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Gregory Piazza, MD, MS, Associate Director, Thrombosis Research Group, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 2018P001681
Record Dates: First submitted 2018-11-01; First posted 2018-11-02 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Chronic Thromboembolic Pulmonary Hypertension
Keywords: echocardiography; pulmonary embolism; pulmonary hypertension; screening
MeSH Terms: conditions — Pulmonary Embolism; Hypertension, Pulmonary

STUDY DESIGN:
Intervention Model Description: 400-patient single-center Quality Improvement Initiative in the form of a randomized controlled trial
Who Masked: Participant
Masking Description: The allocation ratio will be 1:1 for an EPIC BPA on-screen alert versus no notification. Investigators will be assessing the impact of the EPIC BPA on echocardiographic screening for CTEPH and the diagnosis of CTEPH in the patients enrolled in this Quality Improvement Initiative. While investigators will randomize patients by Attending Physician of Record to minimize cluster-effect, the observational unit will be the patient. The cluster-effect describes a type of confounding observed in studies of provider behavior that can result in a bias of the outcome toward the null. In such a case, a provider may carry over knowledge gained from the alert for the intervention group patient to the care of the control group patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alert (Experimental): On-screen computerized decision support alert during the outpatient clinical encounter that notifies the provider that the patient should be screened for CTEPH
  Interventions: Behavioral: On-screen computerized decision support alert
- No Alert (No Intervention): No provider notification

INTERVENTIONS:
Behavioral: On-screen computerized decision support alert — On-screen electronic alert during the outpatient clinical encounter that notifies him or her that the patient should be screened for CTEPH
  Arms: Alert

SUMMARY:
To address the knowledge gap that exists among providers resulting in underdiagnosis of chronic thromboembolic pulmonary hypertension (CTEPH), the investigators have devised this 400-patient single-center Quality Improvement Initiative in the form of a randomized controlled trial of an EPIC Best Practice Advisory (BPA) on-screen alert versus no notification to increase echocardiographic screening for CTEPH and the diagnosis of CTEPH in patients with prior pulmonary embolism (PE) and symptoms/signs suggestive of pulmonary hypertension or recent pulmonary testing suggesting unexplained respiratory symptoms at 3 months.

Aim #1: To determine the impact of a Best Practice Advisory (BPA), using the EPIC Electronic Health Record computerized decision support (CDS) software, on echocardiographic screening for CTEPH in patient with prior PE and symptoms/signs suggestive of pulmonary hypertension or recent pulmonary testing suggesting unexplained respiratory symptoms.

Aim #2: To determine the impact of an EPIC BPA on the diagnosis of CTEPH in patient with prior PE and symptoms/signs suggestive of pulmonary hypertension or recent pulmonary testing suggesting unexplained respiratory symptoms.

DETAILED DESCRIPTION:
Study design: 400-patient single-center Quality Improvement Initiative in the form of a randomized controlled trial. The allocation ratio will be 1:1 for an EPIC Best Practice Advisory (BPA) on-screen alert versus no notification. Investigators will be assessing the impact of the EPIC BPA on echocardiographic screening for chronic thromboembolic pulmonary hypertension (CTEPH) and the diagnosis of CTEPH in the patients enrolled in this Quality Improvement Initiative. While investigators will randomize patients by Attending Physician of Record to minimize cluster-effect, the observational unit will be the patient.

Type of control : The control group will have no electronic alert notification issued to the responsible provider.

Number of subjects: 400 subjects will be enrolled with 200 subjects to be randomized to the alert group and 200 subjects to the control group in a 1:1 allocation ratio.

Primary Efficacy Outcome: Frequency of echocardiographic screening for CTEPH in patients with prior pulmonary embolism (PE) and symptoms/signs suggestive of pulmonary hypertension or recent pulmonary testing suggesting unexplained respiratory symptoms at 3 months. Investigators will review the order entry and cardiology test results sections of the Electronic Health Record (EPIC) to make this determination.

Secondary Efficacy Outcome: Frequency of CTEPH diagnosis at 3 months. The diagnosis of CTEPH will be confirmed by clinical notation in the EHR or a mean pulmonary-artery pressure greater than 25 mmHg that persists 6 months after PE diagnosis.

Safety Outcomes: Because there is no reasonable expectation for adverse events or patient safety concerns with this Quality Improvement Initiative focused on increasing provider awareness about the risk of CTEPH and the indication for screening with echocardiography, investigators will not collect any safety outcomes or variables.

Plan for statistical analysis: The primary statistical analysis will be the comparison of the frequency of echocardiographic screening for CTEPH in the alert group compared with the control (no alert) group. A secondary statistical analysis will be the comparison of the frequency of CTEPH diagnosis in the alert group compared with the control (no alert) group.

ELIGIBILITY:
Inclusion Criteria:

* BWH outpatient
* At least 18 years of age
* Evaluated in Primary Care or Cardiovascular Medicine Clinic
* Persistent or new symptoms/signs suggestive of pulmonary hypertension [syncope, malaise and fatigue, dyspnea, exercise intolerance, hemoptysis, chest pain, dizziness/vertigo, gait abnormality, cardiomegaly, ascites, and peripheral edema] OR recent pulmonary testing (pulmonary function tests [PFTs], chest X-ray, or chest CT) suggesting unexplained respiratory symptoms at least 6 months from the diagnosis of PE
* Have not undergone echocardiography within the prior 6 months

Exclusion Criteria:

* Absence of persistent or new symptoms/signs suggestive of pulmonary hypertension OR recent pulmonary testing (pulmonary function tests [PFTs], chest X-ray, or chest CT) suggesting unexplained respiratory symptoms
* PE within the last 6 months
* Echocardiogram or invasive hemodynamic assessment with the prior 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Frequency of echocardiographic screening for CTEPH in patients with prior PE and symptoms/signs suggestive of pulmonary hypertension or recent pulmonary testing suggesting unexplained respiratory symptoms at 3 months following randomization. | 3 Months
  Investigators will review the Provider Order Entry and cardiology test results sections of the Electronic Health Record (EPIC) to make this determination.

SECONDARY OUTCOMES:
Frequency of CTEPH diagnosis at three months. | 3 Months
  The diagnosis of CTEPH will be confirmed by clinical notation in the EHR or a mean pulmonary artery pressure greater than 25 mmHg that persists 6 months after PE diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Piazza, MD, MS, Principal Investigator — BWH
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Piazza G, Goldhaber SZ. Chronic thromboembolic pulmonary hypertension. N Engl J Med. 2011 Jan 27;364(4):351-60. doi: 10.1056/NEJMra0910203. No abstract available. PMID 21268727